CLINICAL TRIAL: NCT01764282
Title: A Cluster-randomized Controlled Trial of Promoting Antiretroviral Therapy Among Serodiscordant Couples to Reduce HIV Transmission
Brief Title: Promoting Antiretroviral Therapy Among Serodiscordant Couples to Reduce HIV Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012ZX10001007-001
Record Dates: First submitted 2012-12-26; First posted 2013-01-09 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: HIV
Keywords: HIV; serodiscordant couples HIV sero-conversion; anti-retroviral therapy; intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): comprehensive intervention components
  Interventions: Behavioral: comprehensive intervention components
- Usual (No Intervention): According the National HIV Antiretroviral treatment Guideline, provide treatment referrals for those treatment-eligible HIV-positive patients.

INTERVENTIONS:
Behavioral: comprehensive intervention components — ART promotion, Couple testing and consulting promotion, and Condom use promotion
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of reducing HIV transmission among sero-discordant couples by applying comprehensive intervention components.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was carried out in forty counties from 16 cities. The strategy of Social Marketing was applied to influence sero-discordant couples' behavioral changes including safer sexual intercourses, regular HIV testing for the negative partners, antiretroviral therapy initiation.

ELIGIBILITY:
Inclusion Criteria:

* Couples are required to have a stable relationship and live together in the last 3 months;
* Older than 18 years and younger than 60 years; without regard to CD4 count;
* Open cohort(any newly diagnosed serodiscordant couples who are eligible for treatment will be included during the study period).

Exclusion Criteria:

* Couples are not have a stable relationship or do not live together in the last 3 months;
* Younger than 18 years old.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11096 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
HIV seroconversion rate of HIV negatives among HIV serodiscordant couples | up to 2 years

SECONDARY OUTCOMES:
Proportion of HIV positives receiving ART among HIV serodiscordant couples | up to 2 years
The incidence rate of AIDS-related diseases of HIV positives among serodiscordant couples | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zuyou Wu, MD, PHD, Principal Investigator — National Center for AIDS/STD Control and Prevention, China CDC
Locations (5):
- China (5):
  - Center for Disease Control and Prevention,Guangxi Zhuang Autonomous Region, Nanning, Guilin, Laibin, Qinzhou, Guangxi
  - Center for Disease Control and Prevention, Henan Province, Zhumadian, Henan
  - Center for Disease Control and Prevention, Sichuan Province, Liangshan, Sichuan
  - Center for Disease Control and Prevention, Xinjiang Uygur Autonomous Region, Urumchi, Ili, Xinjiang
  - Center for Disease Control and Prevention, Yunnan Province, Kunming, Dehong, Wenshan, Honghe, Yunnan

REFERENCES:
- [Result] Zhang F, Dou Z, Ma Y, Zhang Y, Zhao Y, Zhao D, Zhou S, Bulterys M, Zhu H, Chen RY. Effect of earlier initiation of antiretroviral treatment and increased treatment coverage on HIV-related mortality in China: a national observational cohort study. Lancet Infect Dis. 2011 Jul;11(7):516-24. doi: 10.1016/S1473-3099(11)70097-4. PMID 21600849
- [Result] Cohen MS, Gay CL. Treatment to prevent transmission of HIV-1. Clin Infect Dis. 2010 May 15;50 Suppl 3(0 3):S85-95. doi: 10.1086/651478. PMID 20397961
- [Result] Stephenson R, Barker J, Cramer R, Hall MA, Karita E, Chomba E, Vwalika C, Allen S. The demographic profile of sero-discordant couples enrolled in clinical research in Rwanda and Zambia. AIDS Care. 2008 Mar;20(3):395-405. doi: 10.1080/09540120701593497. PMID 18351489
- [Result] He N, Duan S, Ding Y, Rou K, McGoogan JM, Jia M, Yang Y, Wang J, Montaner JS, Wu Z; China National HIV Prevention Study Group. Antiretroviral therapy reduces HIV transmission in discordant couples in rural Yunnan, China. PLoS One. 2013 Nov 13;8(11):e77981. doi: 10.1371/journal.pone.0077981. eCollection 2013. PMID 24236010